CLINICAL TRIAL: NCT05833490
Title: The Effect of Peripheral Sensory Priming Using Repetitive Peripheral Magnetic Stimulation (rPMS) on Motor Skill Performance in Persons With a Stroke.
Brief Title: The Effect of rPMS on Motor Skill Performance in Persons With a Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0600
Record Dates: First submitted 2023-04-10; First posted 2023-04-27 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: rPMS; motor skill performance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will be blind to the experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sensory-based priming (Experimental): Participants will receive rPMS at 10% above motor threshold with the coil placed on the Tibialis Anterior muscle belly. rPMS parameters will be: 40 trains, intermittently (3) seconds on, (19) seconds off, with an intensity ~10% above motor threshold.
  Interventions: Other: Repetitive Peripheral Magnetic Stimulation (rPMS)
- Sham Priming (Sham Comparator): Participants will receive sham rPMS at a very low intensity with the coil placed on the dorsal part of the foot. rPMS parameters will be: 40 trains, intermittently (3) seconds on, (19) seconds off, with an intensity at 5% of maximum stimulator output.
  Interventions: Other: Sham Priming

INTERVENTIONS:
Other: Repetitive Peripheral Magnetic Stimulation (rPMS) — Repetitive Peripheral Magnetic Stimulation (rPMS) is an external device that delivers repetitive pulsed magnetic fields of sufficient magnitude, will be applied on the tibialis anterior muscle belly at ~ 10% of motor threshold, in order to induce neural action potentials in the lower extremities.
  Arms: Sensory-based priming
Other: Sham Priming — Sham Priming using the Repetitive Peripheral Magnetic Stimulation (rPMS), it will be applied on the dorsal part of the foot with a minimal intensity at 5% of maximum stimulator output, that is of insufficient magnitude to induce changes in the muscle or nerves of lower extremities.
  Arms: Sham Priming

SUMMARY:
In the past two decades, even as stroke cases increase around the world, advances in motor rehabilitation have been limited. Clinical trials of stroke rehabilitation have examined the therapeutic utility of several neuromodulatory devices to improve efficacy of motor training. However, there is limited knowledge on the effects of sensory-based priming techniques using repetitive peripheral magnetic stimulation (rPMS) post stroke. This project focuses on understanding the effect of rPMS on motor skill performance in persons with stroke.

DETAILED DESCRIPTION:
The central hypothesis of this study is that rPMS is a suitable priming technique for enhancing motor skill performance in individuals with stroke. The investigators plan to test our hypothesis by pursuing the following specific aim:

To determine whether rPMS can facilitate lower limb's motor skill performance more than sham rPMS in individuals with stroke.

Hypothesis: The effect of stimulation on lower limb's motor skill performance will be measured using a visuomotor tracking task at different time points: baseline, immediately after, at 30 minutes, and 60 minutes after stimulation. Individuals with stroke during the rPMS condition will demonstrate greater motor skill performance following rPMS and will be able to sustain the enhanced performance at 30 and 60 minutes after the stimulation, compared to sham condition.

This study will improve our understanding of the effects of rPMS, thus encouraging the use of a single session of rPMS as a priming tool to enhance motor skill performance. The proposal is important as it is the first to study the time course effects of rPMS on lower limb's motor skill performance in stroke populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed mono-hemispheric stroke
* More than 3 months since stroke onset.
* Participants must demonstrate adequate cognitive abilities to be able to follow the protocol (21>MMSE).

Exclusion Criteria:

* Individuals with lesions affecting the brainstem or cerebellum.
* Other musculoskeletal or neurological impairments such as (Alzheimer, Parkinson, etc.).
* Complete paralysis that would limit the participant's' ability to perform motor skill tasks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Motor skill performance | at baseline
  The investigators will assess motor skill performance by asking the participants to track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Each trial lasts for 60 seconds. Participants will be asked to perform 10 familiarization trials, this only to make participants familiar with the task. After the familiarization, participants will perform 5 trials at baseline.
Motor skill performance | 0 minutes after the stimulation
  The investigators will assess motor skill performance by asking the participants to track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Each trial lasts for 60 seconds. Participants will be asked to perform 5 trials immediately after the stimulation
Motor skill performance | 30 minutes after the stimulation
  The investigators will assess motor skill performance by asking the participants to track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Each trial lasts for 60 seconds. Participants will be asked to perform 5 trials at 30 minutes after the stimulation
Motor skill performance | 60 minutes after the stimulation
  The investigators will assess motor skill performance by asking the participants to track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Each trial lasts for 60 seconds. Participants will be asked to perform 5 trials at 60 minutes after the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Brain Plasticity lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No